CLINICAL TRIAL: NCT00219817
Title: Safety and Efficacy of RC-1291 HCl in Patients With Cancer Related Anorexia and Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC-1291-203
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Cancer Cachexia
Keywords: Anorexia; Cachexia
MeSH Terms: conditions — Anorexia; Cachexia

INTERVENTIONS:
Drug: RC-1291 HCl

SUMMARY:
Anorexia and weight loss are devastating complications in late-stage cancer patients and is strongly associated with mortality in these patients. Activation of Ghrelin receptors have been demonstrated to stimulate appetite. RC-1291 HCl, by virtue of its ghrelin like activity and Growth Hormone releasing effects may have a dual role in the reversal of cancer induced anorexia and weight loss. This study will test the safety and efficacy of RC-1291 in the treatment of cancer patients with anorexia and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling patients ≥ 18 years of age with incurable, histologically diagnosed cancer.
* Involuntary loss of body weight of ≥ 5 % within the past 6 months

Exclusion Criteria:

* Presently hospitalized or in a nursing care facility.
* Inability to increase food intake from secondary causes.
* Liver disease
* If female-pregnant, breast-feeding or of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Body Weight
Lean Body Mass
Functional Performance

CONTACTS AND LOCATIONS:
Overall Officials: William Polvino, MD, Study Director — Sapphire Therapeutics
Locations (7):
- United States (7):
  - California Cancer Care Center, Greenbrae, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Cancer Outreach Associates, Abingdon, Virginia

REFERENCES:
- [Derived] Garcia JM, Boccia RV, Graham CD, Yan Y, Duus EM, Allen S, Friend J. Anamorelin for patients with cancer cachexia: an integrated analysis of two phase 2, randomised, placebo-controlled, double-blind trials. Lancet Oncol. 2015 Jan;16(1):108-16. doi: 10.1016/S1470-2045(14)71154-4. Epub 2014 Dec 16. PMID 25524795